CLINICAL TRIAL: NCT01632332
Title: A Phase I Trial of the Safety and Immunogenicity of a Multi-epitope HER-2/Neu Peptide Vaccine in Subjects Previously Treated for HER-2 Positive Breast Cancer
Brief Title: Vaccine Therapy in Treating Patients With Previously Treated Stage II-III HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Marker Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1136; NCI-2012-00963 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: HER2-positive Breast Cancer; Male Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (HER-2/neu peptide vaccine) (Experimental): Patients receive HER-2/neu peptide vaccine ID every 28 days for up to 6 courses in the absence of disease recurrence or unacceptable toxicity.
  Interventions: Biological: HER-2/neu peptide vaccine; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: HER-2/neu peptide vaccine — Given ID
  Other Names: HER-2
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The purpose of this study is to look at the safety and immune response to a vaccine used in patients previously treated for HER2 (human epidermal growth factor receptor 2) positive breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile of a peptide-based vaccine targeting HER-2/neu, in patients with stage II/III HER-2 positive breast cancer.

II. To determine the ability of this vaccination protocol to elicit an immune response as measured by activated HER-2/neu-specific T lymphocytes or high-affinity antibodies.

SECONDARY OBJECTIVES:

I. To compile descriptive follow-up data regarding vital status and disease recurrence.

II. To determine if HER-2/neu peptide 885 generates a T cell response that is specific to HER-2/neu or is cross-reactive with epidermal growth factor receptor (EGFR) protein.

III. To determine if the human leukocyte antigen (HLA)-DR epitopes contain HLA class I embedded epitopes.

OUTLINE:

Patients receive HER-2/neu peptide vaccine intradermally (ID) every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 2 additional years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of primary breast cancer, stage II or III, completely resected; Note: history of a local recurrence allowable if also completely resected
* Prior diagnosis of HER-2 positive primary breast cancer using American Society of Clinical Oncologists (ASCO)/College of American Pathologists (CAP) guidelines (either by evidence of 3+ immunohistochemical staining or with in situ hybridization [FISH] amplification)
* Completion of surgery +/- radiation at least 30 days prior to registration
* Must have received mastectomy or lumpectomy plus radiation
* Must have received either neoadjuvant and/or adjuvant chemotherapy for treatment of breast cancer
* Must have received either neoadjuvant and/or adjuvant trastuzumab for treatment of breast cancer
* All chemotherapy, trastuzumab, and/or corticosteroids must be completed at least 90 days prior to registration; Note: hormonal therapy and bisphosphonates may be ongoing
* Clinically without any evidence of disease recurrence/progression (per practice guidelines for breast cancer)
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 75,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Creatinine =< 2 x upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2 x ULN
* Albumin >= 3 g/dL
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Capable of understanding the investigative nature, potential risks, and benefits of the study
* Capable of providing valid informed consent
* Willing to return to enrolling institution (Mayo Clinic Rochester) for all study visits (immunizations, blood draws, etc)
* Willing to employ adequate contraception from the time of registration through 6 months after the final vaccine cycle; Note: adequate contraception methods include birth control pills, barrier device, intrauterine device
* Willing to provide blood samples for correlative research purposes
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Willing to receive a tetanus vaccination if you have not had one within the past year

Exclusion Criteria:

Any prior lapatinib or pertuzumab treatment

Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

* Pregnant women
* Nursing women unwilling to stop breast feeding
* Men or women of child bearing potential who are unwilling to employ adequate contraception from the time of registration through 6 months after the final vaccine cycle Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens Immunocompromised patients including patients known to be human immunodeficiency virus (HIV) positive or those on chronic steroids; Note: must be off systemic steroids at least 90 days prior to registration; topical steroids or steroid eye drops are permitted Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Uncontrolled acute or chronic medical conditions including, but not limited to the following:

* Active infection requiring antibiotics
* Congestive heart failure with New York Heart Association class III or IV; moderate to severe objective evidence of cardiovascular disease
* Myocardial infarction or stroke within previous 6 months Receiving any other investigational agent Other active malignancy at time of registration or within the last three years prior to registration; EXCEPTIONS: non-melanoma skin cancer or carcinoma-in-situ (eg of cervix, prostate); NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment (cytotoxics, monoclonal antibodies, small molecule inhibitors) for their cancer Known history of autoimmune disease, including Type I diabetes Any prior hypersensitivity or adverse reaction to granulocyte-macrophage colony-stimulating factor (GM-CSF) History of trastuzumab-related cardiac toxicity requiring interruption or discontinuation of therapy, even if left ventricular ejection fraction (LVEF) fully recovered Baseline LVEF with a value below 55% Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment History of myocardial infarction =< 168 days (6 months) prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias Bilateral invasive breast cancer, either synchronous or metachronous; Note: ductal carcinoma in situ in the contralateral breast is permissible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-07-09 (Actual); Primary Completion 2014-03-24 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience toxicities of attribution during the course of treatment (grades 3-5 of the NCI's Cancer Therapy Evaluation Program [CTEP] Common Terminology Criteria for Adverse Events, version 4.0) for 2 years. | Assessed up to 2 years following final immunization
  The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
To determine the ability of this vaccination protocol to elicit an immune response as measured by activated HER-2/neu-specific T lymphocytes or high-affinity antibodies | 30 months
  Immune responses to to the vaccine components will be periodically assessed using various assays measuring cytokine release, frequency of T cells, and antibody generation.

SECONDARY OUTCOMES:
Disease-free survival | 30 months
  Disease-free survival is defined as the time from registration to documentation of disease recurrence, second primary, or death without disease recurrence or second primary. The distribution of disease-free and overall survival times will be estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Knutson, Ph.D., Principal Investigator — Mayo Clinic; Amy Degnim, M.D., Principal Investigator — Mayo Clinic; Kimberly Kalli, Ph.D., Study Chair — Mayo Clinic; Timothy Hobday, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States